CLINICAL TRIAL: NCT07375056
Title: The Effect of Therapeutic Play and Virtual Reality Glasses on Pain and Dental Anxiety Before Local Anesthesia in Children: A Randomized Controlled Trial
Brief Title: Effect of Therapeutic Play and Virtual Reality Glasses on Pain and Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehpare Yener, DDS, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-ETHICS-2023-03-07
Record Dates: First submitted 2025-12-29; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety; Pain
Keywords: Therapeutic play; Virtual reality glasses; Local anesthesia; Pediatric dentistry
MeSH Terms: conditions — Pain | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Therapeutic Play Group (Active Comparator): Therapeutic play intervention before local anesthesia
  Interventions: Device: Intervention 1: Therapeutic Play Group
- Arm 2: Virtual Reality Glasses Group (Active Comparator): Use of virtual reality glasses before local anesthesia
  Interventions: Behavioral: Intervention 2: Virtual Reality Glasses Group
- Arm 3: Control Group (Active Comparator): Routine local anesthesia without preparatory intervention
  Interventions: Other: control group

INTERVENTIONS:
Device: Intervention 1: Therapeutic Play Group — Therapeutic play intervention before local anesthesia
  Arms: Arm 1: Therapeutic Play Group
Behavioral: Intervention 2: Virtual Reality Glasses Group — Use of virtual reality glasses before local anesthesia
  Arms: Arm 2: Virtual Reality Glasses Group
Other: control group — Routine local anesthesia without preparatory intervention
  Arms: Arm 3: Control Group

SUMMARY:
Background: A child's first dental experience plays a crucial role in treatment success and in fostering cooperation during future visits. In pediatric dentistry, various non-pharmacological approaches have been implemented to prepare children for dental procedures. This study aims to evaluate the effects of two such approaches-therapeutic play and virtual reality glasses-designed to familiarize children with dental instruments, on pain perception and dental anxiety.

Methods: A total of 66 healthy children aged 6-9 years attending their first dental visit at the Pediatric Dentistry Clinic of Ataturk University will be included. Participants will be randomly assigned into three groups: one group will receive therapeutic play before local anesthesia; the second group will use virtual reality glasses before local anesthesia; and the control group will receive local anesthesia without any preparatory intervention. Dental anxiety and pain will be assessed using the Modified Children's Dental Anxiety Scale (MCDAS), the Wong-Baker FACES Pain Rating Scale (WBS), and the FLACC scale. Physiological parameters including heart rate and oxygen saturation will be recorded before and after anesthesia.

DETAILED DESCRIPTION:
Children often experience dental anxiety during their first dental visit, particularly before local anesthesia. Non-pharmacological approaches such as therapeutic play and virtual reality distraction may help reduce anxiety and pain perception. This randomized controlled trial compared the effectiveness of therapeutic play and virtual reality glasses with routine care in reducing dental anxiety and pain in children aged 6-9 years. Anxiety was assessed using the Modified Children's Dental Anxiety Scale, pain was evaluated using the Wong-Baker FACES Pain Rating Scale and FLACC scale, and physiological parameters were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 9 years
* Attending their first dental visit
* Participation voluntarily approved by both the child and the parent or legal guardian

Exclusion Criteria:

* Presence of acute dental pain
* Presence of systemic health problems
* Allergy to the modeling compound used in the playset
* Any visual or auditory impairment that could interfere with the use of virtual reality glasses

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Dental anxiety score measured by the Modified Child Dental Anxiety Scale (MCDAS) | Baseline (before intervention), Pre-anesthesia (before local anesthesia), Immediately after local anesthesia injection
  Dental anxiety assessed using the Modified Child Dental Anxiety Scale (MCDAS), a validated questionnaire consisting of 8 items. Total scores range from 8 to 40, with higher scores indicating higher dental anxiety.
Pain score measured by the Wong-Baker FACES Pain Rating Scale | Baseline (before intervention), Pre-anesthesia (before local anesthesia), Immediately after local anesthesia injection
  Pain intensity assessed using the Wong-Baker FACES Pain Rating Scale, with scores ranging from 0 to 10, where higher scores indicate more severe pain.
Pain score measured by the FLACC scale | Baseline (before intervention), Pre-anesthesia (before local anesthesia), Immediately after local anesthesia injection
  Pain intensity assessed using the FLACC scale (Face, Legs, Activity, Cry, Consolability), with scores ranging from 0 to 10, where higher scores indicate more severe pain.

SECONDARY OUTCOMES:
Heart Rate (beats per minute) | Pre-anesthesia (before local anesthesia), Immediately after local anesthesia injection
  Heart rate measured using a pulse oximeter
Oxygen Saturation (SpO₂) | Pre-anesthesia (before local anesthesia), Immediately after local anesthesia injection
  Oxygen saturation (SpO₂, %) measured using a pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Mehpare yener, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Faculty of Dentistry, Erzurum, Turkey, Erzurum, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajeswari SR, Chandrasekhar R, Vinay C, Uloopi KS, RojaRamya KS, Ramesh MV. Effectiveness of Cognitive Behavioral Play Therapy and Audiovisual Distraction for Management of Preoperative Anxiety in Children. Int J Clin Pediatr Dent. 2019;12(5):419-22.